CLINICAL TRIAL: NCT06166745
Title: A Prospective, Randomized, Clinical Trial Comparing the Efficacy of Sensi-IP Toothpaste With a Sodium Fluoride Toothpaste in the Treatment of Dentinal Hypersensitivity
Brief Title: Efficacy of Sensi-IP Toothpaste in the Treatment of Dentinal Hypersensitivity Compared to a Sodium Fluoride Toothpaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IR Scientific Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIP001
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Dentinal Hypersensitivity
Keywords: Fluoride; Dentine Hypersensitivity; Toothpaste
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Sensi-IP toothpaste (Experimental): Sodium Fluoride Toothpaste with Sensi-IP
  Interventions: Device: Sensi-IP toothpaste
- Sodium fluoride toothpaste (Active Comparator): Sodium Fluoride Toothpaste
  Interventions: Device: Sodium Fluoride Toothpaste

INTERVENTIONS:
Device: Sensi-IP toothpaste — Brushing daily with the Sensi-IP toothpaste for 14 days for dentinal hypersensitivity.
  Arms: Sensi-IP toothpaste
Device: Sodium Fluoride Toothpaste — Brushing daily with the Sodium Fluoride toothpaste for 14 days for dentinal hypersensitivity.
  Arms: Sodium fluoride toothpaste

SUMMARY:
The study is designed as a prospective, randomized, parallel arm, double blinded, pilot clinical trial.The primary objective is to evaluate the efficacy of Sensi-IP +NaF as compared to a NaF toothpaste in the reduction of dentin hypersensitivity in adult participants over 14 days. Study endpoints include Evaporative Air blast Stimuli (Schiff Airblast Sensitivity Score), Tactile Stimuli (Yeaple probe Assessment), Visual Analogue Scale Evaporative Stimuli and the occurrence of adverse events. The study will include 2 study arms: 1. Sodium fluoride toothpaste with Sensi IP (N=23) and 2. Sodium fluoride toothpaste (N=23). Total of 46 participants (ages 18-80 years) with at least one hypersensitive tooth in 2 different quadrants which are anterior to the molars will be enrolled.

DETAILED DESCRIPTION:
The Study design is a prospective, randomized, parallel arm, double blinded, single study site, proof of concept clinical trial. The study will include 2 study arms: 1) Brushing with sodium fluoride toothpaste with Sensi IP (N=23) and 2) Brushing with sodium fluoride toothpaste (N=23).

A total of 46 adults (18 - 80 years of age) will be included in this clinical trial. To account for the potential of a 15% drop out, as many as 46 participants may be enrolled and treated with the goal of 20 participants per arm.

Study procedures will take place at the following timelines shown below:

Visit 1: Screening Visit -Informed consent; Screening for eligibility

Visit 2: Baseline Day 1: 7 days post screening; (+/- 1 Day) -Confirm eligibility, 1st treatment with allocated product

Visit 3 Day 2: 1 Day after Visit 2; (+1 Day) -Study Assessments

Visit 4: Day 14 (14 days after Visit 2 ;+/ 2 Days) -Final Study Assessments and Study Exit

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to abide by the terms of the consent form
* Can independently sign informed consent
* Participants 18-80 years old
* Agree to abstain from any other desensitizing, (stannous fluoride, arginine, calcium phosphosilicate, nanohydroxy apatite, potassium nitrate and varieties) whitening or other dental procedures for the duration of the trial
* Agree to refrain from all oral hygiene procedures (in addition to the Study Product) and chewing gum for 8 h prior to each scheduled visit and refrained from eating and drinking for 4 h prior to each visit (sips of water is allowed for taking routine medications).
* Have at least two hypersensitive teeth (≥2 Schiff Airblast Sensitivity Score) consistent at screening and baseline.

Target Teeth:

1. Demonstrate cervical dentin exposure, which may be visible with the use of loupes
2. Are non-adjacent in 2 different quadrants, anterior to the molars.

Exclusion Criteria:

* Are pregnant (to be confirmed by an over-the-counter dipstick pregnancy test) or breast feeding
* Have lip or tongue piercing which the subject is unwilling to remove for the duration of the study
* Have an active oral ulcer (Aphthous ulcer) at the time of screening
* Have undergone desensitizing treatment (stannous fluoride, arginine, calcium phosphosilicate, nanohydroxy apatite, potassium nitrate and varieties) within the 1 month preceding the screening visit
* Have undergone tooth bleaching within 8 weeks of screening
* Have undergone scale, polish, interventional dental procedures within 1 month of screening
* Are currently undergoing orthodontics
* Receiving concomitant medication/therapy that might affect dentine hypersensitivity, e.g., regular use (>3X per week) of analgesics, antihistamines, non-steroidal anti-inflammatory drug, and selective serotonin reuptake inhibitor medication
* Demonstrate severe bruxism as indicated by reported muscular pain
* Reduced salivary flow as determined by clinical assessment and/or patient report, diagnosed with Sjogren's disease, received radiation therapy to the head or neck within a year or currently being on medications that may cause xerostomia
* Have generalized gingivitis or active periodontal disease as determined by the clinical exam or undergoing treatment for the above disease
* Have had gingival surgery in the previous six months
* Have allergies to any Study toothpaste ingredients, including the flavor components
* With active caries or any condition such as pulpitis that would precipitate mouth pain
* Who have self-reported eating disorders, uncontrolled gastroesophageal reflux disease (GERD or Acid Reflux), excessive dietary or environmental exposure to acids, or other systemic conditions that are predisposing to dentinal hypersensitivity
* Participated in other clinical trials in the previous 28 days
* Have smoked/vaped or used marijuana in the previous 12 months
* Are diagnosed with unstable mental illness or chronic pain (e.g., fibromyalgia, TMD, migraine, etc.) that could alter the Participant's ability to report pain accurately
* In the opinion of the Investigator, are unable to comply fully with the trial requirements

Target Teeth With:

1. Extensive or unsatisfactory restorations fractures, periodontal alterations, caries lesions, orthodontic brackets, endodontic treatments, or pulp alterations interfering confounding evaluations
2. Crowns, veneers, or bridges

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline at Day 14 using the Schiff Airblast Sensitivity Score | 14 Days
  Schiff Airblast sensitivity score is mainly used to assess participant response to evaporated air stimuli. The scale is 0-3 and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change from baseline at Day 14 using the Yeaple probe assessment | 14 Days
  Dentin Hypersensitivity in response to tactile stimulus is to be determined by Yeaple probe. Teeth were evaluated by stroking the probe across the buccal surface at the cementoenamel junction, perpendicular to the tooth. The preset force exerted by the probe initially was set to 10 gram and was increased progressively in 10-gram increments up to 70 grams or until the patient first reported experiencing discomfort. Higher scores mean a better outcome.
Change from baseline at Day 14 using the Visual Analogue Score (VAS) for pain following evaporative stimuli | 14 Days
  Participants response to evaporative stimuli will be measured by asking participants to rate their pain from zero to 10 (using a 10 cm scale). Higher scores mean worse outcome.

OTHER OUTCOMES:
The occurrence of adverse events that are possibly, probably, or definitely related to the product | 14 days
  Safety will be evaluated by assessing adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Doucette, Study Director — IR Scientific Inc.
Locations (1):
- The Forsyth Institute, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Richmond NL. Dental hypersensitivity: recent advances in diagnosis and treatment. J Indiana Dent Assoc. 1993 Jan-Feb;72(1):20-2. PMID 8478751
- [Background] Davari A, Ataei E, Assarzadeh H. Dentin hypersensitivity: etiology, diagnosis and treatment; a literature review. J Dent (Shiraz). 2013 Sep;14(3):136-45. PMID 24724135
- [Background] Addy M, West NX. The role of toothpaste in the aetiology and treatment of dentine hypersensitivity. Monogr Oral Sci. 2013;23:75-87. doi: 10.1159/000350477. Epub 2013 Jun 28. PMID 23817061
- [Background] Poulsen S, Errboe M, Hovgaard O, Worthington HW. Potassium nitrate toothpaste for dentine hypersensitivity. Cochrane Database Syst Rev. 2001;(2):CD001476. doi: 10.1002/14651858.CD001476. PMID 11405992
- [Background] Mantzourani M, Sharma D. Dentine sensitivity: past, present and future. J Dent. 2013 Jul;41 Suppl 4:S3-17. doi: 10.1016/S0300-5712(13)70002-2. PMID 23929643
- [Background] Shearer A, Montazerian M, Sly JJ, Hill RG, Mauro JC. Trends and perspectives on the commercialization of bioactive glasses. Acta Biomater. 2023 Apr 1;160:14-31. doi: 10.1016/j.actbio.2023.02.020. Epub 2023 Feb 16. PMID 36804821
- [Background] Hu ML, Zheng G, Zhang YD, Yan X, Li XC, Lin H. Effect of desensitizing toothpastes on dentine hypersensitivity: A systematic review and meta-analysis. J Dent. 2018 Aug;75:12-21. doi: 10.1016/j.jdent.2018.05.012. Epub 2018 May 19. PMID 29787782
- [Background] MacDonald K, Boudreau E, Thomas GV, Badrock TC, Davies LJ, Lloyd MJ, Spradbery PS, Turner-Cahill S, Boyd D. In vitro evaluation of Sensi-IP(R): A soluble and mineralizing sensitivity solution. Heliyon. 2021 Dec 25;8(1):e08672. doi: 10.1016/j.heliyon.2021.e08672. eCollection 2022 Jan. PMID 35036593
- [Background] Bakri MM, Hossain MZ, Razak FA, Saqina ZH, Misroni AA, Ab-Murat N, Kitagawa J, Saub RB. Dentinal tubules occluded by bioactive glass-containing toothpaste exhibit high resistance toward acidic soft drink challenge. Aust Dent J. 2017 Jun;62(2):186-191. doi: 10.1111/adj.12484. Epub 2017 May 22. PMID 27813093
- [Background] Schiff T, Delgado E, Zhang YP, Cummins D, DeVizio W, Mateo LR. Clinical evaluation of the efficacy of an in-office desensitizing paste containing 8% arginine and calcium carbonate in providing instant and lasting relief of dentin hypersensitivity. Am J Dent. 2009 Mar;22 Spec No A:8A-15A. PMID 19472556
- [Background] Nathoo S, Delgado E, Zhang YP, DeVizio W, Cummins D, Mateo LR. Comparing the efficacy in providing instant relief of dentin hypersensitivity of a new toothpaste containing 8.0% arginine, calcium carbonate, and 1450 ppm fluoride relative to a benchmark desensitizing toothpaste containing 2% potassium ion and 1450 ppm fluoride, and to a control toothpaste with 1450 ppm fluoride: a three-day clinical study in New Jersey, USA. J Clin Dent. 2009;20(4):123-30. PMID 19831165
- [Background] Seong J, Newcombe RG, Foskett HL, Davies M, West NX. A randomised controlled trial to compare the efficacy of an aluminium lactate/potassium nitrate/hydroxylapatite toothpaste with a control toothpaste for the prevention of dentine hypersensitivity. J Dent. 2021 May;108:103619. doi: 10.1016/j.jdent.2021.103619. Epub 2021 Feb 26. PMID 33647373
- [Derived] Hasturk H, Boyd D, MacDonald-Parsons K, Turner-Cahill S, Seong J, West N, Doucette HJ. Comparative efficacy of novel bioactive glass versus sodium fluoride toothpaste for dentin hypersensitivity. J Periodontol. 2025 Dec 10. doi: 10.1002/jper.70024. Online ahead of print. PMID 41373067